CLINICAL TRIAL: NCT04237324
Title: A Prospective, Randomized Controlled Split-face Trial of a Fractional Microneedle Radiofrequency Device（FMR） and Fractional Erbium-Doped Glass 1,565-nm Device(NAFL) Therapy in Baggy Lower Eyelids
Brief Title: Efficacy of Fractional Microneedle Radiofrequency and Fractional Erbium-Doped Glass 1,565-nm for Baggy Lower Eyelids
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: No.KY20172045-C-1
Record Dates: First submitted 2019-12-24; First posted 2020-01-23 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2019-11

CONDITIONS: Photoaging

STUDY DESIGN:
Intervention Model Description: The purpose of this study is to assess the safety and efficacy of FMR and NAFL for the treatment of BLEs in Asian. After being informed about the study and potential risks, all patients giving written informed consent. Patients were randomly divided into FMR side and NAFL opposite side 3 times in total at a 1-month interval. FMR side has been used by FMR device (INFINI, Lutronic Co., Goyang-si, Korea) and the NAFL side has been used by ResurFX module of M22 (Lumenis Co., Yokneam, Israel).
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NAFL group (Experimental): One side of the patient face has been therapied by 1565nm fiber nonablative fractional laser(Lumenis Co., Yokneam, Israel).
  Interventions: Procedure: Treatment one side BLE by NAFL
- FMR group (Active Comparator): Another side of the patient face has been therapied by FMR device (INFINI, Lutronic Co., Goyang-si, Korea).
  Interventions: Procedure: Treatment another side BLE by FMR

INTERVENTIONS:
Procedure: Treatment one side BLE by NAFL — One side of the patient face underwent treatment using the ResurFX module of M22 (Lumenis Co., Yokneam, Israel) randomly.
  Arms: NAFL group
Procedure: Treatment another side BLE by FMR — One side of the patient face underwent treatment using FMR device (INFINI, Lutronic Co., Goyang-si, Korea).
  Arms: FMR group

SUMMARY:
The purpose of this study was to compare the efficacy and safety of FMR and NAFL in the treatment of baggy lower eyelids(BLEs)

DETAILED DESCRIPTION:
Fifteen baggy lower eyelids(BLEs) volunteers were recruited prospectively. Everyone was divided into two groups with FMR and NAFL according to the random number table. One side of the face was treated with FMR device and the other side was treated with NAFL device. Subjective and objective adverse reactions were recorded during the operation. Subjective adverse reactions were recorded after each treatment. The VAS score of patient satisfaction and the blind method score of standard photo observer were used for subjective evaluation, and the objective evaluation was carried out by using VISIA，Antera-3D and CineScan.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Bags lower eyelids ( BLEs )；
2. Two senior attending surgeons diagnosed the BLEs;
3. The clinical diagnosis standard was mild swelling or puffiness under the eyes;
4. Between 18 to 60 years old.

Exclusion Criteria:

1. History of retinoic acid;
2. History of hormone use;
3. History of keloids;
4. History of injection of botulinum toxin or filler at the site of treatment;
5. Skin inflammation or facial infection;
6. Pregnancy or lactation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction Scores(PSS) | Change from Baseline PSS at 1-month after 3rd treatment, Change from Baseline PSS at 3-month after 3rd treatment, Change from 1-month after 3rd treatment PSS at 3-month after 3rd treatment.
  Patients scored their satisfaction used 10-point Visual analogue scales (VAS, 0 = unsatisfied, 10= very satisfied)
Blinded Investigator Assesement(BIA) | Change from Baseline BIA at 1-month after 3rd treatment, Change from Baseline BIA at 3-month after 3rd treatment, Change from 1-month after 3rd treatment BIA at 3-month after 3rd treatment.
  The physician's severity score of standard photographs used VAS 0-4(VAS, 0 = no eyelid bags, 4= very obvious eyelid bags)
Periorbital wrinkles assessment by VISIA system(VISIA) | Change from Baseline VISIA at 1-month after 3rd treatment, Change from Baseline VISIA at 3-month after 3rd treatment, Change from 1-month after 3rd treatment VISIA at 3-month after 3rd treatment.
  VISIA Complexion Analysis System (Canfield Imaging Systems, Fairfield, New Jersey, USA)
Change of BLEs by ANTERA-3D(ANTERA-3D) | Change from Baseline ANTERA-3D at 1-month after 3rd treatment, Change from Baseline ANTERA-3D at 3-month after 3rd treatment, Change from 1-month after 3rd treatment ANTERA-3D at 3-month after 3rd treatment.
  volume of elevations (mm3), elevation area (mm2), and the maximum peak height volume of elevations (mm3), elevation area (mm2), and the maximum peak height We assessment the volume(mm3), elevation area (mm2), and the maximum peak height (mm) of elevations(mm) by ANRERA-3D camera (Miravex Limited, Ireland).
Orbital fat depth and length by CineScan assessment(CineScan) | Change from Baseline CineScan at 1-month after 3rd treatment, Change from Baseline CineScan at 3-month after 3rd treatment, Change from 1-month after 3rd treatment CineScan at 3-month after 3rd treatment.
  Orbital fat depth(mm) and length(mm) by CineScan Ultrasonic Ophthalmic A and B scan System (Quantel Medical Inc., Bozeman, Montana, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Xianjie Ma, Ph.D, Principal Investigator — Department of Plastic Surgery,Xijing Hospital
Locations (1):
- Department of Plastic Surgery, Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared for patient privacy

REFERENCES:
- [Result] Sachs ME, Bosniak SL. Correction of true periorbital fat herniation in cosmetic lower lid blepharoplasty. Aesthetic Plast Surg. 1986;10(2):111-4. doi: 10.1007/BF01575278. PMID 3526832
- [Result] Camirand A, Doucet J, Harris J. Anatomy, pathophysiology, and prevention of senile enophthalmia and associated herniated lower eyelid fat pads. Plast Reconstr Surg. 1997 Nov;100(6):1535-46. doi: 10.1097/00006534-199711000-00026. PMID 9385969
- [Result] Goldberg RA, McCann JD, Fiaschetti D, Ben Simon GJ. What causes eyelid bags? Analysis of 114 consecutive patients. Plast Reconstr Surg. 2005 Apr 15;115(5):1395-402; discussion 1403-4. doi: 10.1097/01.prs.0000157016.49072.61. PMID 15809605
- [Result] Castanares S. Classification of baggy eyelids deformity. Plast Reconstr Surg. 1977 May;59(5):629-33. No abstract available. PMID 850700
- [Result] Zarem HA, Resnick JI. Expanded applications for transconjunctival lower lid blepharoplasty. Plast Reconstr Surg. 1991 Aug;88(2):215-20; discussion 221. PMID 1852813
- [Result] Roberts TL 3rd. Laser blepharoplasty and laser resurfacing of the periorbital area. Clin Plast Surg. 1998 Jan;25(1):95-108. PMID 9507800
- [Result] Roberts TL 3rd, Yokoo KM. In pursuit of optimal periorbital rejuvenation: laser resurfacing with or without blepharoplasty and brow lift. Aesthet Surg J. 1998 Sep-Oct;18(5):321-32. doi: 10.1016/s1090-820x(98)70086-x. PMID 19328157
- [Result] Beylot C, Grognard C, Michaud T. [Ablative and fractional lasers]. Ann Dermatol Venereol. 2009 Oct;136 Suppl 6:S311-9. doi: 10.1016/S0151-9638(09)72539-6. French. PMID 19931691
- [Result] Jordan R, Cummins C, Burls A. Laser resurfacing of the skin for the improvement of facial acne scarring: a systematic review of the evidence. Br J Dermatol. 2000 Mar;142(3):413-23. doi: 10.1046/j.1365-2133.2000.03350.x. PMID 10735944
- [Result] Manstein D, Herron GS, Sink RK, Tanner H, Anderson RR. Fractional photothermolysis: a new concept for cutaneous remodeling using microscopic patterns of thermal injury. Lasers Surg Med. 2004;34(5):426-38. doi: 10.1002/lsm.20048. PMID 15216537
- [Result] Kaplan H, Kaplan L. Combination of microneedle radiofrequency (RF), fractional RF skin resurfacing and multi-source non-ablative skin tightening for minimal-downtime, full-face skin rejuvenation. J Cosmet Laser Ther. 2016 Dec;18(8):438-441. doi: 10.1080/14764172.2016.1228981. Epub 2016 Oct 5. PMID 27594273
- [Result] Gershonowitz A, Gat A. VoluDerm microneedle technology for skin treatments-in vivo histological evidence. J Cosmet Laser Ther. 2015 Feb;17(1):9-14. doi: 10.3109/14764172.2014.957219. Epub 2014 Sep 25. PMID 25151912
- [Result] Lee HJ, Seo SR, Yoon MS, Song JY, Lee EY, Lee SE. Microneedle fractional radiofrequency increases epidermal hyaluronan and reverses age-related epidermal dysfunction. Lasers Surg Med. 2016 Feb;48(2):140-9. doi: 10.1002/lsm.22420. Epub 2015 Sep 28. PMID 26415023
- [Result] Tanaka Y. Long-term three-dimensional volumetric assessment of skin tightening using a sharply tapered non-insulated microneedle radiofrequency applicator with novel fractionated pulse mode in asians. Lasers Surg Med. 2015 Oct;47(8):626-33. doi: 10.1002/lsm.22401. Epub 2015 Aug 14. PMID 26272454
- [Result] Manuskiatti W, Pattanaprichakul P, Inthasotti S, Sitthinamsuwan P, Hanamornroongruang S, Wanitphakdeedecha R, Chu-Ongsakol S. Thermal Response of In Vivo Human Skin to Fractional Radiofrequency Microneedle Device. Biomed Res Int. 2016;2016:6939018. doi: 10.1155/2016/6939018. Epub 2016 May 9. PMID 27247943
- [Result] Seo KY, Yoon MS, Kim DH, Lee HJ. Skin rejuvenation by microneedle fractional radiofrequency treatment in Asian skin; clinical and histological analysis. Lasers Surg Med. 2012 Oct;44(8):631-6. doi: 10.1002/lsm.22071. Epub 2012 Aug 30. PMID 22936274
- [Result] Harth Y, Frank I. In vivo histological evaluation of non-insulated microneedle radiofrequency applicator with novel fractionated pulse mode. J Drugs Dermatol. 2013 Dec;12(12):1430-3. PMID 24301245
- [Result] Lee SJ, Kim JI, Yang YJ, Nam JH, Kim WS. Treatment of periorbital wrinkles with a novel fractional radiofrequency microneedle system in dark-skinned patients. Dermatol Surg. 2015 May;41(5):615-22. doi: 10.1097/DSS.0000000000000216. PMID 25899885
- [Result] Jeon IK, Chang SE, Park GH, Roh MR. Comparison of microneedle fractional radiofrequency therapy with intradermal botulinum toxin a injection for periorbital rejuvenation. Dermatology. 2013;227(4):367-72. doi: 10.1159/000356162. Epub 2013 Nov 21. PMID 24280617
- [Result] McCrudden MT, McAlister E, Courtenay AJ, Gonzalez-Vazquez P, Singh TR, Donnelly RF. Microneedle applications in improving skin appearance. Exp Dermatol. 2015 Aug;24(8):561-6. doi: 10.1111/exd.12723. Epub 2015 May 26. PMID 25865925
- [Result] Seo KY, Kim DH, Lee SE, Yoon MS, Lee HJ. Skin rejuvenation by microneedle fractional radiofrequency and a human stem cell conditioned medium in Asian skin: a randomized controlled investigator blinded split-face study. J Cosmet Laser Ther. 2013 Feb;15(1):25-33. doi: 10.3109/14764172.2012.748201. PMID 23368685 (Retraction: PMID 33739221 J Cosmet Laser Ther. 2020 Jul 3;22(4-5):215)
- [Result] Naouri M, Mazer JM. Non-insulated microneedle fractional radiofrequency for the treatment of scars and photoaging. J Eur Acad Dermatol Venereol. 2016 Mar;30(3):499-502. doi: 10.1111/jdv.12890. Epub 2015 Jan 5. No abstract available. PMID 25560082
- [Result] Hantash BM, Ubeid AA, Chang H, Kafi R, Renton B. Bipolar fractional radiofrequency treatment induces neoelastogenesis and neocollagenesis. Lasers Surg Med. 2009 Jan;41(1):1-9. doi: 10.1002/lsm.20731. PMID 19143021
- [Result] Polder KD, Bruce S. Radiofrequency: Thermage. Facial Plast Surg Clin North Am. 2011 May;19(2):347-59. doi: 10.1016/j.fsc.2011.04.006. PMID 21763995
- [Result] Chae WS, Seong JY, Jung HN, Kong SH, Kim MH, Suh HS, Choi YS. Comparative study on efficacy and safety of 1550 nm Er:Glass fractional laser and fractional radiofrequency microneedle device for facial atrophic acne scar. J Cosmet Dermatol. 2015 Jun;14(2):100-6. doi: 10.1111/jocd.12139. Epub 2015 Mar 23. PMID 25810322
- [Result] Fitzpatrick R, Geronemus R, Goldberg D, Kaminer M, Kilmer S, Ruiz-Esparza J. Multicenter study of noninvasive radiofrequency for periorbital tissue tightening. Lasers Surg Med. 2003;33(4):232-42. doi: 10.1002/lsm.10225. PMID 14571447
- [Result] Guertler A, Reinholz M, Steckmeier S, Gauglitz GG. Evaluation of a non-ablative, fractional 1565 nm laser for the improvement of striae distensae albae. J Eur Acad Dermatol Venereol. 2019 Jan;33(1):220-226. doi: 10.1111/jdv.15228. Epub 2018 Oct 8. PMID 30169914
- [Result] Yang S, Kim BR, Kim HS, Choi CW, Jo SJ, Youn SW. A quantitative, objective method for evaluating the surgical outcomes of baggy eyelid correction using orbital gray scale analysis. J Cosmet Dermatol. 2019 Dec;18(6):1814-1820. doi: 10.1111/jocd.12922. Epub 2019 Mar 20. PMID 30895705
- [Result] Guertler A, Reinholz M, Poetschke J, Steckmeier S, Schwaiger H, Gauglitz GG. Objective evaluation of the efficacy of a non-ablative fractional 1565 nm laser for the treatment of deliberate self-harm scars. Lasers Med Sci. 2018 Feb;33(2):241-250. doi: 10.1007/s10103-017-2348-x. Epub 2017 Oct 27. PMID 29080008
- [Result] Linming F, Wei H, Anqi L, Yuanyu C, Heng X, Sushmita P, Yiming L, Li L. Comparison of two skin imaging analysis instruments: The VISIA(R) from Canfield vs the ANTERA 3D(R) CS from Miravex. Skin Res Technol. 2018 Feb;24(1):3-8. doi: 10.1111/srt.12381. Epub 2017 Jun 5. PMID 28585335
- [Derived] Dou W, Yang Q, Yin Y, Fan X, Qiu L, Yang Z, Jian Z, Song W, Ma X. A randomized, split-face controlled trial on the safety and effects of microneedle fractional radiofrequency and fractional erbium-doped glass 1,565-nm laser therapies for baggy lower eyelids. J Cosmet Laser Ther. 2021 Aug;23(5-6):105-112. doi: 10.1080/14764172.2021.2001532. Epub 2021 Nov 23. PMID 34812096

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-12-08): https://cdn.clinicaltrials.gov/large-docs/24/NCT04237324/Prot_SAP_000.pdf
  • Informed Consent Form (2017-12-08): https://cdn.clinicaltrials.gov/large-docs/24/NCT04237324/ICF_001.pdf